CLINICAL TRIAL: NCT04758936
Title: Effect of Clonidine vs. Dexmedetomidine in Addition to Standard Treatment in Agitated Delirium in Intensive Care Patients: Pilot Study.
Brief Title: Clonidine vs. Dexmedetomidine in Agitated Delirium in Intensive Care Patients
Acronym: Clodex
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Olivier Lheureux, MD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2020/421
Record Dates: First submitted 2021-02-10; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Delirium; Critical Illness
Keywords: Clonidine; Dexmedetomidine; Delirium; intensive care
MeSH Terms: conditions — Delirium; Critical Illness | interventions — Clonidine; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clonidine (Experimental): Given that agitated delirium requires rapid medical intervention, α-2 agonist therapy (clonidine) will be administered as soon as possible, The sedative and analgesic treatments will be administered and titrated according to the scales on the usual protocol of the service (evaluation of sedation (NICS) and analgesia (VAS, BPS, BPS-NI). In case of excessive sedation assessed by the scores and administration of combined treatments (α-2 agonist and other sedatives), the reduction of the doses of other sedatives will be preferred over the α-2 agonist treatment. In case of insufficient sedation despite maximal doses of α-2 agonist, other sedatives (choosen by the attending physician) will administered and titrated according to the scales for pain and sedation evaluation.
  Interventions: Drug: Clonidine
- Dexmedetomidine (Experimental): Given that agitated delirium requires rapid medical intervention, α-2 agonist therapy (dexmedetomidine) will be administered as soon as possible. The α-2 agonist treatment that will be started will depend on the allocation of the previously randomized unit. The sedative and analgesic treatments will be administered and titrated according to the scales on the usual protocol of the service (evaluation of sedation (NICS) and analgesia (VAS, BPS, BPS-NI). In case of excessive sedation assessed by the scores and administration of combined treatments (α-2 agonist and other sedatives), the reduction of the doses of other sedatives will be preferred over the α-2 agonist treatment. In case of insufficient sedation despite maximal doses of α-2 agonist, other sedatives (choosen by the attending physician) will administered and titrated according to the scales for pain and sedation evaluation.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Clonidine — The doses administered (clonidine 1500mg diluted in NaCl0.9% solution of 50 ml) ranged from 0.01μg/kg/min to 0.03μg/kg/min.
  Other Names: Dexmedetomidine
  Arms: Clonidine
Drug: Dexmedetomidine — The doses administered (dexmedetomidine 200mg diluted in NaCl0.9% 50ml) ranged from 0.4μg/kg/h and can be titrated up to 1.4μg/kg/h.
  Arms: Dexmedetomidine

SUMMARY:
Delirium is one of the most common manifestations of cerebral dysfunction in severely ill patients.

The international guidelines for the prevention of delirium in intensive care recommend the daily application of environmental, behavioral and pharmacological strategies. In the case of the agitated form of delirium, experts recommend the use of low-dose neuroleptics and α-2 agonists to control psychotic manifestations rather than traditional sedatives (mainly benzodiazepines) that can clearly aggravate delirium.

Currently, two pharmacological α-2 agonists, clonidine (Catapressan®, Boehringer Ingelheim) and dexmedetomidine (Dexdor®, Orion Corporation), are marketed and commonly used in intensive care for their sedative, anxiolytic and analgesic properties.

To our knowledge, no studies have compared the effects of clonidine and dexmedetomidine in agitated delirium in intensive care patients. Therefore, our goal is to compare the safety of clonidine and dexmedetomidine (in terms of bradycardia and / or hypotension) in addition to standard treatment in the context of agitated delirium in intensive care patients.

DETAILED DESCRIPTION:
Delirium is one of the most common manifestations of cerebral dysfunction in severely ill patients (60 to 80% of ventilated patients), leading not only to short-term complications (prolonged duration of ventilation, prolonged hospital stay, and increased mortality) but also long-term repercussions in the form of impaired cognitive functions, post-traumatic stress syndromes, and decreased quality of life. Different forms of delirium coexist: some patients are very agitated while others are, on the contrary, in an apathetic state. In intensive care patients, the agitated form of delirium is particularly problematic because of the risk of self-extubation and removal of other critical medical devices.

Pain, stress, anxiety and deregulation of wake / sleep cycles are important risk factors for delirium occurrence and are unfortunately frequently encountered in varying degrees in intensive care.

The international guidelines for the prevention of delirium in intensive care recommend the daily application of environmental, behavioral and pharmacological strategies. Thus, the early mobilization of the patient, the respect of the waking / sleep cycles, the adequate control of the pain represent effective measures of prevention. These guidelines also emphasize the importance of minimal use of sedative treatments while ensuring the comfort and safety of patients.

Finally, in the case of the agitated form of delirium, experts recommend the use of low-dose neuroleptics and α-2 agonists to control psychotic manifestations rather than traditional sedatives (mainly benzodiazepines) that can clearly aggravate delirium.

The α-2 receptors constitute a family of receptors coupled to transmembrane G proteins with 3 pharmacological subtypes, α-2A, α-2B and α-2C. The α-2A and α-2C subtypes are mainly found in the central nervous system. Stimulation of these receptor subtypes may be responsible for sedation, analgesia and sympatholytic effects. Α-2B receptors are more common on vascular smooth muscle and have been shown to have vasopressor effects. By their inhibitory action on adenylyl cyclase, the 3 subtypes have several effects: 1) they reduce the levels of cyclic adenosine monophosphate, 2) they cause a hyperpolarization of noradrenergic neurons in the brain stem, in particular in the locus ceruleus, 3) they suppress the neural discharge. This suppression inhibits the release of norepinephrine into the synapse resulting in a modulatory effect on the anxiety, wakefulness and sleep of patients. Activation of this negative feedback loop may also result in reduced heart rate and blood pressure by sympatholytic action.

Currently, two pharmacological α-2 agonists, clonidine (Catapressan®, Boehringer Ingelheim) and dexmedetomidine (Dexdor®, Orion Corporation), are marketed and commonly used in intensive care for their sedative, anxiolytic and analgesic properties. Unlike traditional sedatives (benzodiazepines and propofol) that leave the patient unresponsive to stimuli or stupor, sedation achieved by administering these α-2 agonists has several advantages. The α-2 agonists lower the general level of alertness (NREM, indifference to the environment and pain), but leave the waking ability intact. Therefore, under α-2 agonists, patients are more easily awake until a return to full consciousness, able to respond to simple orders, participate in their sessions of physiotherapy and communicate, within the limits of the presence of an intubation probe or non-invasive ventilation mask. In addition, these agents do not cause respiratory depression.

Clonidine is an α-2 agonist that has an affinity of 200/1 for α-2 receptors versus α-1 receptors. Initially marketed for its antihypertensive properties, clonidine is used in intensive care for its sedative and analgesic effects, especially in the treatment of delirium or alcohol withdrawal syndromes (alcohol, opioids, or benzodiazepines). The pharmacodynamics of this α-2 agonist is characterized by hepatic metabolism and renal elimination. The half-life elimination time is about 24 hours. The doses administered ranged from 0.01 μg / kg / min to 0.03 μg / kg / min and the main reported side effects were: bradycardia, low blood pressure and dry mouth. Pharmacodynamically, clonidine has the advantage to be very affordable (about 90 euros per patient for a week of treatment).

Dexmedetomidine is the newest of the α-2 agonists. Its affinity and specificity for α-2 receptors is much greater than that of clonidine (1600/1 α-2 / α-1 receptors)25. The pharmacodynamics of this α-2 agonist is characterized by hepatic metabolism and elimination almost completely renal. The half-life elimination time is about 2 hours. The recommended doses vary between 0.4 μg / kg / h and can be titrated up to 1.4 μg / kg / h. The main reported side effects are: bradycardia and low blood pressure. Its cost, on the other hand, is much higher (800 euros per patient for a one week treatment). The efficacy of dexmedetomidine has been demonstrated in terms of reduced mechanical ventilation time and ICU length of hospitalization when compared to placebo, traditional sedatives (propofol or benzodiazepines), neuroletics in the context of critical care delirium.

To date, only one study has compared the effects of clonidine and dexmedetomidine in a prospective, randomized manner (n = 70) in order to achieve short-term deep sedation in post-operative mechanical ventilation patients. Study confirms sedative efficacy of α-2 agonists and suggests greater hemodynamic stability under dexmedetomidine.

To our knowledge, no studies have compared the effects of clonidine and dexmedetomidine in agitated delirium in intensive care patients. Therefore, our goal is to compare the safety of clonidine and dexmedetomidine (in terms of bradycardia and / or hypotension) in addition to standard treatment in the context of agitated delirium in intensive care patients. Bradycardia is defined by a heart rate <60 / min (or a decrease of 20% of the initial heart rate) and arterial hypotension by one of the following criteria:

* systolic blood pressure less than 90mmHg o(r a decrease of 20% of the initial systolic arterial pressure)
* initiation of a vasopressor treatment
* 10% increase in the dose of vasopressor treatment, if already started

ELIGIBILITY:
Inclusion Criteria:

* present agitated delirium, confirmed by the CAM-ICU diagnostic scale
* require mechanical restraint or psychotropic / sedative

Exclusion Criteria:

* Acute neurological central or medullary problems (vascular, traumatic, infectious, tumoral causes)
* Severe hepatic insufficiency (Child C cirrhosis)
* Severe renal insufficiency (creatinine clearance <30ml / min) or renal replacement therapy
* Bradycardia <60 / min
* 2nd or 3rd degree atrioventricular block (unless placed pacemaker)
* Hemodynamic instability (MAP <60mmHg despite adequate vascular filling and vasopressor treatment).
* Pregnant woman or breastfeeding
* Use of α-2 agonist or antagonist agents within 24 hours of randomization
* Allergy known to one of the α-2 agonists used in the study
* Moribund patient (survival prognosis at limited 24h or therapeutic de-escalation envisaged)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
hemodynamic tolerance | Up to 7 days
  Bradycardia is defined by a heart rate <60 / min (or a decrease of 20% of the initial heart rate) and arterial hypotension by one of the following criteria:
  * systolic blood pressure less than 90mmHg o(r a decrease of 20% of the initial systolic arterial pressure)
  * initiation of a vasopressor treatment
  * 10% increase in the dose of vasopressor treatment, if already started

SECONDARY OUTCOMES:
number of living days without ventilation over 28 days | Up to 28 days
time to obtain a sedative sedation score (NICS -1 to 1) | up to 7 days
  NICS = Nursing instrument confusion score. From -3 to + 3. Positive means agitation. Negative means sedation.
time to obtain a first CAM-ICU test indicating the absence of delirium | Up to 7 days
  Confusion assessment method in ICU). CAM ICU positive means delirium.
duration of delirium by evaluation CAM-ICU | Up to 7 days
  Confusion assessment method in ICU). CAM ICU positive means delirium.
use of other sedative and psychotropic medications (number and total doses) | Up to 7 days
number of catheters / agitation extubation | Up to 7 days
Number of patients with tracheostomy | Up to 28 days
daily assessment of organ dysfunction by SOFA score | Up to 7 days
  Sequential Organ Failure assessment score. From 0 to 24. 24 means worse outcome.
28 day survival or exit from the ICU | Up to 28 days
length of stay USI | through study completion, an average of 2 years
length of hospital stay | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Creteur Jacques, MD PhD, Study Director — CUB Erasme Hospital ULB
Locations (3):
- Belgium (3):
  - CUB Erasme Hospital ULB, Brussels
  - Civil hospital Marie Curie, Charleroi
  - Clinique Saint-Pierre, Ottignies

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] van den Boogaard M, Schoonhoven L, Evers AW, van der Hoeven JG, van Achterberg T, Pickkers P. Delirium in critically ill patients: impact on long-term health-related quality of life and cognitive functioning. Crit Care Med. 2012 Jan;40(1):112-8. doi: 10.1097/CCM.0b013e31822e9fc9. PMID 21926597
- [Background] Girard TD, Pandharipande PP, Ely EW. Delirium in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S3. doi: 10.1186/cc6149. Epub 2008 May 14. PMID 18495054
- [Background] Dubois MJ, Bergeron N, Dumont M, Dial S, Skrobik Y. Delirium in an intensive care unit: a study of risk factors. Intensive Care Med. 2001 Aug;27(8):1297-304. doi: 10.1007/s001340101017. PMID 11511942
- [Background] Reade MC, Finfer S. Sedation and delirium in the intensive care unit. N Engl J Med. 2014 Jan 30;370(5):444-54. doi: 10.1056/NEJMra1208705. No abstract available. PMID 24476433
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] DAS-Taskforce 2015; Baron R, Binder A, Biniek R, Braune S, Buerkle H, Dall P, Demirakca S, Eckardt R, Eggers V, Eichler I, Fietze I, Freys S, Frund A, Garten L, Gohrbandt B, Harth I, Hartl W, Heppner HJ, Horter J, Huth R, Janssens U, Jungk C, Kaeuper KM, Kessler P, Kleinschmidt S, Kochanek M, Kumpf M, Meiser A, Mueller A, Orth M, Putensen C, Roth B, Schaefer M, Schaefers R, Schellongowski P, Schindler M, Schmitt R, Scholz J, Schroeder S, Schwarzmann G, Spies C, Stingele R, Tonner P, Trieschmann U, Tryba M, Wappler F, Waydhas C, Weiss B, Weisshaar G. Evidence and consensus based guideline for the management of delirium, analgesia, and sedation in intensive care medicine. Revision 2015 (DAS-Guideline 2015) - short version. Ger Med Sci. 2015 Nov 12;13:Doc19. doi: 10.3205/000223. eCollection 2015. PMID 26609286
- [Background] Buerkle H, Yaksh TL. Pharmacological evidence for different alpha 2-adrenergic receptor sites mediating analgesia and sedation in the rat. Br J Anaesth. 1998 Aug;81(2):208-15. doi: 10.1093/bja/81.2.208. PMID 9813525
- [Background] Pichot C, Ghignone M, Quintin L. Dexmedetomidine and clonidine: from second- to first-line sedative agents in the critical care setting? J Intensive Care Med. 2012 Jul-Aug;27(4):219-37. doi: 10.1177/0885066610396815. Epub 2011 Apr 27. PMID 21525113
- [Background] Patel SB, Kress JP. Sedation and analgesia in the mechanically ventilated patient. Am J Respir Crit Care Med. 2012 Mar 1;185(5):486-97. doi: 10.1164/rccm.201102-0273CI. Epub 2011 Oct 20. PMID 22016443
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the Intensive Care Unit: executive summary. Am J Health Syst Pharm. 2013 Jan 1;70(1):53-8. doi: 10.1093/ajhp/70.1.53. PMID 23261901
- [Background] Miyazaki S, Uchida S, Mukai J, Nishihara K. Clonidine effects on all-night human sleep: opposite action of low- and medium-dose clonidine on human NREM-REM sleep proportion. Psychiatry Clin Neurosci. 2004 Apr;58(2):138-44. doi: 10.1111/j.1440-1819.2003.01207.x. PMID 15009817
- [Background] Huupponen E, Maksimow A, Lapinlampi P, Sarkela M, Saastamoinen A, Snapir A, Scheinin H, Scheinin M, Merilainen P, Himanen SL, Jaaskelainen S. Electroencephalogram spindle activity during dexmedetomidine sedation and physiological sleep. Acta Anaesthesiol Scand. 2008 Feb;52(2):289-94. doi: 10.1111/j.1399-6576.2007.01537.x. Epub 2007 Nov 14. PMID 18005372
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Ruokonen E, Parviainen I, Jakob SM, Nunes S, Kaukonen M, Shepherd ST, Sarapohja T, Bratty JR, Takala J; "Dexmedetomidine for Continuous Sedation" Investigators. Dexmedetomidine versus propofol/midazolam for long-term sedation during mechanical ventilation. Intensive Care Med. 2009 Feb;35(2):282-90. doi: 10.1007/s00134-008-1296-0. Epub 2008 Sep 16. PMID 18795253
- [Background] Martin E, Ramsay G, Mantz J, Sum-Ping ST. The role of the alpha2-adrenoceptor agonist dexmedetomidine in postsurgical sedation in the intensive care unit. J Intensive Care Med. 2003 Jan-Feb;18(1):29-41. doi: 10.1177/0885066602239122. PMID 15189665
- [Background] Hoy SM, Keating GM. Dexmedetomidine: a review of its use for sedation in mechanically ventilated patients in an intensive care setting and for procedural sedation. Drugs. 2011 Jul 30;71(11):1481-501. doi: 10.2165/11207190-000000000-00000. PMID 21812509
- [Background] Venn RM, Hell J, Grounds RM. Respiratory effects of dexmedetomidine in the surgical patient requiring intensive care. Crit Care. 2000;4(5):302-8. doi: 10.1186/cc712. Epub 2000 Jul 31. PMID 11056756
- [Background] Bohrer H, Bach A, Layer M, Werning P. Clonidine as a sedative adjunct in intensive care. Intensive Care Med. 1990;16(4):265-6. doi: 10.1007/BF01705163. PMID 2358560
- [Background] Liatsi D, Tsapas B, Pampori S, Tsagourias M, Pneumatikos I, Matamis D. Respiratory, metabolic and hemodynamic effects of clonidine in ventilated patients presenting with withdrawal syndrome. Intensive Care Med. 2009 Feb;35(2):275-81. doi: 10.1007/s00134-008-1251-0. Epub 2008 Aug 16. PMID 18709354
- [Background] Giovannitti JA Jr, Thoms SM, Crawford JJ. Alpha-2 adrenergic receptor agonists: a review of current clinical applications. Anesth Prog. 2015 Spring;62(1):31-9. doi: 10.2344/0003-3006-62.1.31. PMID 25849473
- [Background] Roberts DJ, Haroon B, Hall RI. Sedation for critically ill or injured adults in the intensive care unit: a shifting paradigm. Drugs. 2012 Oct 1;72(14):1881-916. doi: 10.2165/11636220-000000000-00000. PMID 22950534
- [Background] Gertler R, Brown HC, Mitchell DH, Silvius EN. Dexmedetomidine: a novel sedative-analgesic agent. Proc (Bayl Univ Med Cent). 2001 Jan;14(1):13-21. doi: 10.1080/08998280.2001.11927725. PMID 16369581
- [Background] Yapici N, Coruh T, Kehlibar T, Yapici F, Tarhan A, Can Y, Ozler A, Aykac Z. Dexmedetomidine in cardiac surgery patients who fail extubation and present with a delirium state. Heart Surg Forum. 2011 Apr;14(2):E93-8. doi: 10.1532/HSF98.201011102. PMID 21521683
- [Background] Reade MC, O'Sullivan K, Bates S, Goldsmith D, Ainslie WR, Bellomo R. Dexmedetomidine vs. haloperidol in delirious, agitated, intubated patients: a randomised open-label trial. Crit Care. 2009;13(3):R75. doi: 10.1186/cc7890. Epub 2009 May 19. PMID 19454032
- [Background] Carrasco G, Baeza N, Cabre L, Portillo E, Gimeno G, Manzanedo D, Calizaya M. Dexmedetomidine for the Treatment of Hyperactive Delirium Refractory to Haloperidol in Nonintubated ICU Patients: A Nonrandomized Controlled Trial. Crit Care Med. 2016 Jul;44(7):1295-306. doi: 10.1097/CCM.0000000000001622. PMID 26925523
- [Background] Reade MC, Eastwood GM, Bellomo R, Bailey M, Bersten A, Cheung B, Davies A, Delaney A, Ghosh A, van Haren F, Harley N, Knight D, McGuiness S, Mulder J, O'Donoghue S, Simpson N, Young P; DahLIA Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Effect of Dexmedetomidine Added to Standard Care on Ventilator-Free Time in Patients With Agitated Delirium: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1460-8. doi: 10.1001/jama.2016.2707. PMID 26975647
- [Background] Srivastava U, Sarkar ME, Kumar A, Gupta A, Agarwal A, Singh TK, Badada V, Dwivedi Y. Comparison of clonidine and dexmedetomidine for short-term sedation of intensive care unit patients. Indian J Crit Care Med. 2014 Jul;18(7):431-6. doi: 10.4103/0972-5229.136071. PMID 25097355